CLINICAL TRIAL: NCT04101409
Title: Impact of Shared Decision-Making With Decision Aids on Acoustic Neuroma Treatment Choice: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, tsaiyichieh, Principal Investigator, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: N201711048
Record Dates: First submitted 2019-01-23; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Neuroma, Acoustic
Keywords: decision aids; shared decision making
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAs group (Experimental): Shared decision making using decision aids
  Interventions: Other: Decision aids
- Control group (No Intervention): Standard oral explanation guided with booklets

INTERVENTIONS:
Other: Decision aids — Shared decision making with decision aids
  Arms: DAs group

SUMMARY:
Patients with acoustic neuroma had several treatment options. One of standard treatment is to receive the Gamma knife stereotactic radiosurgery, other options included suboccipital craniotomy and conservative treatment. Thus, shared decision making (SDM) is necessary to aid patients to choose an appropriate treatment that suits their needs.

The investigators have developed a decision aids (DAs) and plan to conduct a randomized controlled trial (RCT) to evaluate its impact on acoustic neuroma patients. The measurements include a battery of interview-based questionnaires and evaluations of decision regret and post-treatment depression. The investigators expect the DAs would benefit the intervention group in the aspects of knowledge, communication and anxiety status during and after their treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acoustic neuroma.
2. Tumor diameter ≤ 3.5cm.
3. The tumor type is Schwannoma.

Exclusion Criteria:

1. Patients with acoustic neuroma less than 20 years old
2. Pregnant woman
3. Patients can not cooperate with Gamma Knife treatment
4. Patients with acoustic neuroma who do not have their own abilities
5. Tumor diameter > 3.5cm.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-02-29 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict | 4 weeks after discussion of treatment choice
  Total score of decisional conflict scale
Knowledge | 4 weeks after discussion of treatment choice
  Total score on knowledge scale

SECONDARY OUTCOMES:
Decision regret | 4 weeks after treatment
  Total score of decision regret, The dependent variable for this study was decision regret, assessed using the Decision Regret Scale (DRS). The DRS consists of five statements: (1) It was the right decision; (2) I regret the choice that was made; (3) I would go for the same choice if I had to do it over again; (4) the choice did me a lot of harm, and (5) the decision was a wise one. Agreement with each statement is measured on a five-point Likert scale (1 = strongly agree to 5 = strongly disagree). Score of each item is converted to a 0-100 scale by subtracting 1 from each item and multiplying by 25. Scores from items 2 and 4 are reversed. To obtain a global score, all items are summed and the total is divided by 5. Scores range from 0 (no regret) to 100 (high regret), increasing by increments of 5.
  Ref. Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D Med Decis Making. 2003 Jul-Aug; 23(4):281-92.
Post-treatment depression | 4 weeks after treatment
  Total score of Hospital anxiety and depression scale (HADS)

IPD SHARING:
Plan to Share IPD: Undecided